CLINICAL TRIAL: NCT06507098
Title: Effectiveness of Telematic Instruction to Patients in the Correct Performance of Respiratory Polygraphy at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Principal Investigator, Alejandro Robles, Head of Pneumology Department, Consorci Sanitari del Maresme
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/23
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-assisted training (Experimental): Patients received a QR code and a link for access to a YouTube video recorded where the process of setting up the respiratory polygraph was explained.
  Interventions: Other: Video-assisted training
- Nurse training (Placebo Comparator): A trained nurse with long experience in home sleep studies explained the setup of the Respiratory Polygraph.
  Interventions: Other: Nurse training

INTERVENTIONS:
Other: Video-assisted training — Patients received a QR code and a link for access to a YouTube video recorded to this effect where the process of setting up the respiratory polygraph was explained. The contents of the video were the same as those in the face-to-face instructions. The visualization of the video was at home, and it could be viewed as many times as necessary.
  Arms: Video-assisted training
Other: Nurse training — A trained nurse with long experience in home sleep studies explained the setup of the respiratory polygraph. At the end of the intervention doubts about the procedure were addressed. Patients did not have access to the video.
  Arms: Nurse training

SUMMARY:
The objective of this trial is to evaluate the use of a video-assisted training for the use of a home-respiratory polygraph for the diagnosis of obstructive sleep apnea compared to standard training by a nurse.

A clinical trial is conducted to this effect. One arm is video-assisted training and the other arm is conventional training by a nurse.

DETAILED DESCRIPTION:
Hypotheses:

1. The use of a video for the correct performance of home respiratory polygraphy (RP) reduces the number of errors derived from poor placement of the polygraph.
2. The degree of satisfaction of telematic instruction will be higher than that of in-person instruction.
3. Telematic instruction will achieve a reduction in care time allocated to instruction for the nursing staff of the Pneumology Day Hospital.

Objectives:

Main objective:

Compare the number of errors in the RP record derived from poor placement of the polygraph between an in-person nursing instruction and a telematic instruction using a video.

Secondary objectives:

* Compare the number of total errors in the RP record between an in-person nursing instruction and a telematic instruction using a popular video.
* Compare the level of patient satisfaction between in-person nursing instruction and telematic instruction using a video.
* Compare the time invested in nursing at the Pneumology Day Hospital in the delivery and instruction of polygraph use between in-person instruction and telematic instruction.

Study design:

Open randomized clinica trial with two arms of intervention: instruction in the functioning of the respiratory polygraph according to usual clinical practice and instruction in audiovisual media.

Study population Patients with suspected Obstructive sleep apnea (OSA) who have been indicated for performing a home respiratory polygraphy for the first time.

Study exhibition Consecutive patients with OSA who come to the Pneumology Service for the collection of a respiratory polygraph for the performance of a home PR for the first time. Recruitment is made at the time you go to collect the respiratory polygraph if you decide to participate in the study, after signing the informed consent and checking the inclusion and exclusion criteria. At that moment randomization will be made and they will be assigned to one of the two intervention groups.

Statistical analysis

The data will be registered in an electronic data base in a dissociated manner so that the analyzers will not be able to connect the identity of the persons participating in the study. The database will be stored in the CSdM information system along with standard security measures. The analysis plan includes:

1. Description of the main characteristics of the study sample (age, gender, participation of a third person, number of views, etc.) including values and typical deviations for numerical variables and percentages for categorical variables.
2. Assessment of the homogeneity and/or comparability of the two study groups. The categorical variables are compared using the Khi al quadrat test or the Fisher exact test and the numerical variables with the T-Student test or the Man Whitney U test.
3. Comparison of the main results measures (percentage of valid PRs, number of errors, satisfaction, investment times) between the two study groups using the same statistical tests as in the previous section.
4. Description of the main causes of error with percentage percentages for each of the identified causes.
5. Evaluation of the factors associated with an invalid RPR using the statistical tests previously carried out and estimating the corresponding OR and the six 95% confidence intervals (95% CI) using bivariate and multivariate logistic regression (to adjust for possible risk factors). confused)
6. Assessment of secondary objects. In all statistical analyses, a statistical significance level of 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age with a clinical suspicion of obstructive sleep apnea who had never undergone respiratory polygraphy

Exclusion Criteria:

* physical, mental or instrumental impairment for video-assisted training;
* the absence of a third person who could collaborate in the setup of the RP;
* the absence of internet connections;
* misunderstanding of Catalan or Spanish languages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Number of valid respiratory polygraphies | 1 day
  Number of studies without recording errors

SECONDARY OUTCOMES:
Personal care time used in the training of the procedure | 1 day
  Minutes of caregiver's time spent in the instruction
Satisfaction with the instruction | 1 day
  Satisfaction of the patients with the instruction measured by an analogic visual scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Robles, MD PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Mateu Serra-Prat, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No